CLINICAL TRIAL: NCT04939389
Title: Comparing a Sensor for Movement Assessment With Traditional Clinical Assessment Methods in Patients After Knee Surgery.
Acronym: MA-KNEE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: crossklinik AG (Other)
Collaborators: Basel Academy for Quality and Research in Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MA-KNEE
Record Dates: First submitted 2021-05-30; First posted 2021-06-25 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2022-07

CONDITIONS: Status After Knee Surgery

STUDY DESIGN:
Intervention Model Description: Paired measurements with two different measurement methods
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Orthelligent Pro — The sensor is attached to the knee of the participant and eight different movement exercises are performed

SUMMARY:
Eight parameters measurable by the sensor "Orthelligent Pro" are compared with traditional measurements based on a goniometer or video taping. The aim is to inform potential users about the distribution of the differences they have to expect when moving from traditional measurement methods to the new sensor.

Patients will perform eight corresponding movement exercises at a single study visit.

DETAILED DESCRIPTION:
In patients suffering from musculo-skeletal disorders, the restoration of full functioning is an important goal of many interventions. Assessment of functioning is often based on corresponding tests. If functioning is related to specific movement patterns, accelerometers and similar sensors are promising to allow a simple and objective assessment, and may replace traditional assessment methods, e.g. based on measurements with the goniometer. Corresponding products tend to enter the market and face clinicians and patients with the question, to which degree they are reliable and comparable with the traditional assessment methods.

Recently, a sensor named "Orthelligent Pro" has been released by the medical device company OPED and is today commercially available. The sensor - to be attached to the knee of a subject - offers the opportunity to assess several parameters related to movement patterns in the lower extremities that are of relevance in the rehabilitation process of orthopedic patients.

The aim of the current project is to inform potential users of this sensor about the difference they have to expect when compared to traditional assessment techniques of the same parameters and about the reproducibility of the measurements both based on the sensor and based on traditional assessments.

Patients of a single clinic will be offered participation. The patients will perform the eight exercises at a single study visit arranged as an addition to a routine follow up visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients after knee surgery (ACL reconstruction, total or partial knee arthroplasty, knee arthroscopy etc.) who are scheduled to a clinical follow up assessment by the surgeon between 4 months and 15 months after surgery.
* Informed consent

Exclusion Criteria:

* Age below 18 years
* Patients who underwent surgery in the lower extremities within the last 4 months
* Patients with severe acute pain
* Patients with contraindications to perform the movements/exercises
* Patients who underwent surgery also at the contralateral leg since the surgery related to the current follow up visit
* Patients who cannot follow the instructions due to language or cognitive problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Tilt angle of the leg in degrees during passive movement of the leg (knee joint) | At the single study visit directly after enrollment of the patient.
Tilt angle of the leg in degrees during active movement of the leg (knee joint) | At the single study visit directly after enrollment of the patient.
Tilt angle of the leg in degrees during leg stretching | At the single study visit directly after enrollment of the patient.
Inward tilt of the lower leg in degrees/on an ordinal assessment scale during one-legged squat | At the single study visit directly after enrollment of the patient.
Angle reproduction when moving the lower leg to three randomly chosen angles | At the single study visit directly after enrollment of the patient.
Jump height at vertical jump (on one leg) | At the single study visit directly after enrollment of the patient.
Inward tilt of the lower leg in degrees/on an ordinal assessment scale at drop jump | At the single study visit directly after enrollment of the patient.
Number of jumps during 30s side hops | At the single study visit directly after enrollment of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Eymann, MSc, Principal Investigator — crossklinik AG
Locations (1):
- crossklinik AG, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available on request
Supporting Information: Study Protocol
Time Frame: The data will become available after publication of the study results

REFERENCES:
- [Result] Eymann J, Vach W, Fischer L, Jakob M, Gosele A. Comparing a Sensor for Movement Assessment with Traditional Physiotherapeutic Assessment Methods in Patients after Knee Surgery-A Method Comparison and Reproducibility Study. Int J Environ Res Public Health. 2022 Dec 9;19(24):16581. doi: 10.3390/ijerph192416581. PMID 36554461